CLINICAL TRIAL: NCT05791812
Title: Application of Direct Current Transcranial stImulation, Remotely superVised in Chronic fATiguE - Heimanwendung Der Transkraniellen Gleichstromstimulation Zur Behandlung Der Chronischen Fatigue
Brief Title: Application of Direct Current Transcranial stImulation, Remotely superVised in Chronic fATiguE
Acronym: ACTIVATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Clinical Professor, MD, Ph.D., University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-3028-101
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Keywords: transcranial direct current stimulation
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- active treatment (Experimental): 2mA of tDCS for 20 min every weekday for six weeks
  Interventions: Device: home-based transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: home-based transcranial direct current stimulation (tDCS) — 2mA of tDCS for 20 min every weekday for six weeks

SUMMARY:
It is a one-arm open-label interventional study with transcranial direct current stimulation in an remote home-based setting with the aims to evaluate the feasibility (usability of the device, compliance of patients, usability of the teletherapy), the effectiveness (clinical ratings) and the compatability of this intervention in 20 patients with myalgic encephalomyelitis/chronic fatigue syndrome.

ELIGIBILITY:
Inclusion Criteria:

* ME/CFS diagnosis according to the Canadian Consensus Criteria
* residence near Regensburg and mother language German
* written informed consent
* stable medication if possible

Exclusion Criteria:

* contraindications for transcranial direct current stimulation
* certain neurological conditions as assessed by study physician
* participation in another study
* pregnancy and lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Usability for the patients | 6 weeks
  Rating of the usability of the treatment (home treatment and video monitoring) with the user experience questionnaire [1-7, 26 items, the higher the better]
Usability for the handlers/clinicians | 6 weeks
  Rating of the usability of the treatment (home treatment and video monitoring) with the user experience questionnaire [1-7, 26 items, the higher the better]
Number of days out of 30 the patients used the device | 6 weeks
  Number of days out of 30 the patients used the device
Number of patients who completed the treatment regularly | 6 weeks
  Number of patients who completed the treatment regularly
Number of responders according the the clinical global impression change score for patients in the per protocol analysis | 6 weeks
  Number of responders according the the clinical global impression change score for patients in the per protocol analysis (range: 1-7; the lower the better)
Effect size for change of fatigue for patients in the per protocol analysis measured with the Bell Score | 6 weeks
  Effect size for change of fatigue for patients in the per protocol analysis measured with the Bell Score (fatigue scale; 0-100; the higher the better)
Effect size for change of fatigue for patients in the per protocol analysis measured with the Chalder Fatigue Scale | 6 weeks
  Effect size for change of fatigue for patients in the per protocol analysis measured with the Chalder Fatigue Scale (fatigue scale; 0-33; the lower the better)

SECONDARY OUTCOMES:
Major Depression Inventory | 18 weeks
  Depression inventory (0-50, the lower the better)
World Health Organisation Quality of life scale (abbreviated Version) (WHOQOL-BREF) | 18 weeks
  Quality of life scale inventory (4-20, the higher the better)
Clinical Global Impression change | 18 weeks
  Clinical Global Impression (1-7, the lower the better)
Pittsburgh sleep quality index | 18 weeks
  sleep inventory (0-21, the lower the better)
numeric analogue scale pain | 18 weeks
  pain scale (0-10, the lower the better)
d2 test | 18 weeks
  concentration test (percentiles; the higher the better)
digital span | 18 weeks
  memory test (percentiles; the higher the better)
Chalder fatigue scale | 18 weeks
  fatigue scale (0-33; the lower the better)
Bell score | 18 weeks
  fatigue scale (0-100; the higher the better)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Principal Investigator — University of Regensburg
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No
On demand possible.